CLINICAL TRIAL: NCT03047369
Title: The Myelin Disorders Biorepository Project and Global Leukodystrophy Initiative Clinical Trials Network
Brief Title: The Myelin Disorders Biorepository Project
Acronym: MDBP
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Biogen (Industry); Eli Lilly and Company (Industry); Myrtelle Inc. (Industry); Orchard Therapeutics Ltd. (Unknown); Passage Bio, Inc. (Industry); Synaptix Biotherapeutics Ltd. (Unknown); Takeda (Industry); Boehringer Ingelheim (Industry); Ionis Pharmaceuticals, Inc. (Industry); Sanofi Winthrop Industrie (Unknown); Sana Biotechnology (Industry); Yaya Foundation for 4H Leukodystrophy (Unknown); University of Pennsylvania (Other); United MSD Foundation (Unknown); Foundation to Fight H-ABC (Unknown); Calliope Joy Foundation (Unknown); Don't Forget Me Foundation (Unknown)
Responsible Party: Principal Investigator, Adeline Vanderver, MD, Program Director, Leukodystrophy Center, Children's Hospital of Philadelphia
Other Study IDs: 14-011236; U54NS115052 (NIH); U01NS106845 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-09 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Leukodystrophy; White Matter Disease; Leukoencephalopathies; 4H Syndrome; Adrenoleukodystrophy; AMN; ALD; ALD Gene Mutation; ALD (Adrenoleukodystrophy); X-linked Adrenoleukodystrophy; X-ALD; Adrenomyeloneuropathy; Aicardi Goutieres Syndrome; AGS; Alexander Disease; Alexanders Leukodystrophy; AxD; ADLD; Canavan Disease; CTX; Cerebrotendinous Xanthomatoses; Krabbe Disease; GALC Deficiency; Globoid Leukodystrophy; TUBB4A-Related Leukodystrophy; H-ABC - Hypomyelination, Atrophy of Basal Ganglia and Cerebellum; HBSL; HBSL - Hypomyelination, Brain Stem, Spinal Cord, Leg Spasticity; LBSL; Leukoencephalopathy With Brain Stem and Spinal Cord Involvement and High Lactate Syndrome (Disorder); Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation; ALSP; CSF1R Gene Mutation; HCC - Hypomyelination and Congenital Cataract; MLC1; Megalencephalic Leukoencephalopathy With Subcortical Cysts; MLD; Metachromatic Leukodystrophy; PMD; Pelizaeus-Merzbacher Disease; PLP1 Null Syndrome; PLP1 Gene Duplication | Blood or Tissue | Mutations; Pelizaeus Merzbacher Like Disease; Peroxisomal Biogenesis Disorder; Zellweger Syndrome; Refsum Disease; Salla Disease; Sialic Storage Disease; Sjögren; Sjogren-Larsson Syndrome; Van Der Knapp Disease; Vanishing White Matter Disease; Charcot-Marie-Tooth; CMT; Mct8 (Slc16A2)-Specific Thyroid Hormone Cell Transporter Deficiency; Allan-Herndon-Dudley Syndrome; Cadasil; Cockayne Syndrome; Multiple Sulfatase Deficiency; Gangliosidoses; GM2 Gangliosidosis; BPAN; Labrune Syndrome; LCC; Mucopolysaccharidoses; TBCK-Related Intellectual Disability Syndrome
Keywords: leukodystrophy; white matter disease; leukoencephalopathy; myelin; demyelinating; mdbp
MeSH Terms: conditions — Leukoencephalopathies; Attention Deficit Disorder with Hyperactivity; Adrenoleukodystrophy; Aicardi-Goutieres syndrome; Alexander Disease; Alexanders leukodystrophy; Canavan Disease; Xanthomatosis, Cerebrotendinous; Leukodystrophy, Globoid Cell; Leukodystrophy, Hypomyelinating, 6; Leukoencephalopathy with Brainstem and Spinal Cord Involvement and Lactate Elevation; Leukodystrophy, Hypomyelinating, 5; Megalencephalic leukoencephalopathy with subcortical cysts; Leukodystrophy, Metachromatic; Pelizaeus-Merzbacher Disease; Peroxisomal Disorders; Zellweger Syndrome; Refsum Disease; Sialic Acid Storage Disease; Sjogren's Syndrome; Sjogren-Larsson Syndrome; Charcot-Marie-Tooth Disease; Allan-Herndon-Dudley syndrome; CADASIL; Cockayne Syndrome; Multiple Sulfatase Deficiency Disease; Gangliosidoses; Gangliosidoses, GM2; Leukoencephalopathy Brain Calcifications and Cysts; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Samples may be collected from affected subjects, as well as healthy controls. Samples may include blood, skin punch biopsy, CSF, urine, etc.) collected either for research or in the context of clinical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Myelin Disorders Biorepository Project (MDBP) seeks to collect and analyze clinical data and biological samples from leukodystrophy patients worldwide to support ongoing and future research projects. The MDBP is one of the world's largest leukodystrophy biorepositories, having enrolled nearly 2,000 affected individuals since it was launched over a decade ago.

Researchers working in the biorepository hope to use these materials to uncover new genetic etiologies for various leukodystrophies, develop biomarkers for use in future clinical trials, and better understand the natural history of these disorders. The knowledge gained from these efforts may help improve the diagnostic tools and treatment options available to patients in the future.

DETAILED DESCRIPTION:
Genetic white matter disorders (leukodystrophies) are estimated to have an incidence of approximately 1:7000 live births. In the past, patients with white matter disease of unknown cause evaluated by the investigator achieved a diagnosis in fewer than 46% of cases after extensive conventional clinical testing. Even when a diagnosis is achieved, the diagnosis takes an average of eight years and this "odyssey" results in testing charges to patients and insurers in excess of $8,000 on average per patient, including patients who never achieve a diagnosis at all. With next generation approaches such as whole exome sequencing, the diagnostic efficacy is closer to 70%, but approximately a third of individuals do not achieve a specific etiologic diagnosis. These diagnostic challenges represent an urgent and unresolved gap in knowledge and disease characterization, as obtaining a definitive diagnosis is of paramount importance for leukodystrophy patients.

Moreover, the mechanisms of disease in many leukodystrophies of known cause are very poorly understood, with little known about the best symptomatic management and, thus, limited standards of care are available for the management of these patients.

The purpose of this study is to: (Aim 1) Define novel homogeneous groups of patients with unclassified leukodystrophy and work toward finding the cause of these disorders; (Aim 2) assess the validity and utility of next-generation sequencing in the diagnosis of leukodystrophies; (Aim 3) establish disease mechanisms in selected known leukodystrophies; (Aim 4) track current care and natural history of these patients to define the longitudinal course and determinants of outcomes in these disorders; (Aim 5) contact subjects for future research studies and/or clinical programs.

This biorepository will use available basic science and clinical research approaches to establish novel diagnoses, biomarkers, and outcome measures for future clinical diagnostic and therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria (Affected Subjects):

* Male or female of any age;
* Suspected or confirmed diagnosis of leukodystrophy or other disorder affecting the white matter of the brain based primarily on the finding of central nervous system neuroimaging consistent with this diagnosis or on an existing diagnosis of a leukodystrophy or genetic leukoencephalopathy as defined in existing classification systems, or in the presence of variant(s) of uncertain significance or genotype consistent with leukodytrophy;
* Documentation of informed consent by the subject, parent, or legal guardian, and, if appropriate, documentation of assent;
* Willingness to provide clinical data, participate in standardized assessments, and/or provide biologic samples.

Exclusion Criteria (Affected Subjects)

* Established diagnosis at the time of referral that is not consistent with a genetic disorder of the white matter, such as an acquired demyelinating condition (e.g. multiple sclerosis), or an infectious etiology, with the exception of sequelae of congenital infections such as CMV;
* Inability to provide consent.

Inclusion Criteria (Healthy Controls)

* Male or female of any age;
* Individuals with no confirmed or suspected diagnosis of leukodystrophy or other disorder affecting the white matter of the brain (including affected patients' caregivers);
* Documentation of informed consent by the subject, parent, or legal guardian, and, if appropriate, documentation of assent.

Exclusion Criteria (Healthy Controls)

- Inability to provide consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Affected subjects will have either a confirmed or suspected diagnosis of leukodystrophy, or a related heritable disorder affecting the white matter of the brain. Healthy controls must be individuals in whom no leukodystrophy or related disorder has been suspected or confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2016-12-08 (Actual); Primary Completion 2030-12-08 (Estimated); Study Completion 2030-12-08 (Estimated)

PRIMARY OUTCOMES:
Define Novel Homogeneous Groups of Patients with Unclassified Leukodystrophy | 10 years from enrollment
  In patients with an unclassified leukodystrophy, the study team will collect as much information as available from existing medical records including existing clinical evaluations, neuropsychological/rehabilitation evaluations, and results from blood, urine, spinal fluid, radiological, and peripheral tissue pathological tests. This data will be evaluated to create nosologic groups amongst patients with unclassified leukodystrophy. Additionally, this aim includes the collection and long-term banking of biological samples in subjects with classified and unclassified leukodystrophies to develop a biorepository. These samples will be compared to samples collected from control subjects, either collected directly from enrolled subjects or through existing banked biological samples.

SECONDARY OUTCOMES:
Assess Validity of Next-Generation Sequencing in the Diagnosis of Leukodystrophies | 10 years from enrollment
  Unclassified leukodystrophy patients enrolled in this study may undergo next generation sequencing approaches, including research whole exome sequencing (WES), whole genome sequencing (WGS), RNA sequencing and high throughput genomics analysis in parallel to standard clinical testing to achieve novel molecular classifications.
Assess Utility of Next-Generation Sequencing in the Diagnosis of Leukodystrophies | 10 years from enrollment
  Clinical utility defined as changes in care and clinical state, included changes in medical morbidities, surgeries, pharmacologic management of complications and implementation of disease specific therapies.
Track Current Care of Leukodystrophy Patients | 10 years from enrollment
  Includes a longitudinal collection of clinical data on diagnostic and therapeutic interventions in leukodystrophy patients and related controls.
Track Natural History of Leukodystrophy Patients | 10 years from enrollment
  Includes longitudinal collection of clinical data on disease presentation, progression and morbidities.
Establish Disease Mechanisms in Leukodystrophies | 10 years from enrollment
  Specific leukodystrophies will be selected for further mechanistic study, using clinical and laboratory tools to establish increased understanding of the underlying pathophysiology. The over-riding hypothesis of this aim is that integrated biochemical, genomic, metabolic, histologic and immunologic profiles of patients with leukodystrophy will define downstream pathway changes consistent with primary defects causing white matter disease. Appropriate controls will be used for comparison to disease related samples.
Contact for Future Research Studies and/or Clinical Programs | 10 years from enrollment
  Individuals enrolled in the study may be informed of other research studies, either at the Children's Hospital of Philadelphia or another site affiliated or not affiliated with this study, that may be of interest to them and/or their their families based on a specific diagnosis or lack thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Vanderver, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (23):
- United States (23):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University (Lucile Packard Children's Hospital), Palo Alto, California
  - University of California, Davis (UC Davis Health), Sacramento, California
  - University of California, San Diego (Rady Children's Hospital), San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University (Children's Healthcare of Atlanta), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine (Texas Children's Hospital), Houston, Texas
  - UT Health Houston, Houston, Texas
  - University of Utah (Primary Children's Hospital), Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to researchers, sponsors, and other stakeholders. Data Use Agreement (DUA) must be put in place with any recipient of IPD. Only aggregate data will be shared publicly.
Time Frame: IPD may be shared at any time.
Access Criteria: Only aggregate data will be shared publicly. Please contact a member of the central study team for information regarding the release of IPD.

REFERENCES:
- [Derived] Adang LA, Schlotawa L, Groeschel S, Kehrer C, Harzer K, Staretz-Chacham O, Silva TO, Schwartz IVD, Gartner J, De Castro M, Costin C, Montgomery EF, Dierks T, Radhakrishnan K, Ahrens-Nicklas RC. Natural history of multiple sulfatase deficiency: Retrospective phenotyping and functional variant analysis to characterize an ultra-rare disease. J Inherit Metab Dis. 2020 Nov;43(6):1298-1309. doi: 10.1002/jimd.12298. Epub 2020 Aug 20. PMID 32749716